CLINICAL TRIAL: NCT03431038
Title: Cross-sectional Study of Prevalence Rate of Abdominal Aortic Aneurysm in OSAHS Patients From BTCH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 17084-0310
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Sleep Apnea, Obstructive; AAA - Abdominal Aortic Aneurysm
MeSH Terms: conditions — Sleep Apnea, Obstructive; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study explore AAA prevalence in OSAHS patients by ultrasound screening and try to analysis risk factors of AAA in OSAHS patients.

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) is an extremely high mortality disease, and ultrasound has been recommended for the screening of AAA, which is highly sensitive and specific. Studies have shown that screening for AAA in the population can significantly reduce deaths from ruptured abdominal aortic aneurysms. However, those study mainly focus on cardiovascular disease patients or general population, no previous study target on obstructive sleep apnea hypopnea syndrome (OSAHS) population. Retrospective studies show that the incidence of apnea syndrome in patients with abdominal aortic aneurysm is higher than that in the control group, which suggests that OSAHS may be one of the causes of abdominal aortic aneurysm. At present, there is no relevant research on the screening of AAA in OSAHS population.

The main objective of this study was to screen the prevalence of AAA in OSAHS population by a cross-sectional study.

ELIGIBILITY:
Inclusion Criteria:

* All patients who accept respiratory sleep monitoring in the department of ENT, BTCH, aged over 45 years, from 2018-01-01 to 2019-12-30

Exclusion Criteria:

* 1. Any previous diagnosis of AAA history;
* 2. Received AAA related treatment;
* 3. Past imaging test result suggested increased diameter of the abdominal aorta.
* 4. Poor compliance; refused to follow the requirements set in this study follow-up, and refused to sign informed consent.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosis as OSAHS
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Diameter of aorta | 0-48 hours
  Diameter of aorta measured by ultrasound

SECONDARY OUTCOMES:
ABI | 0-48 hours
  Ankel brachal index measured by Angiolab 2 - Phlebolab Doppler-System
Carotid artery stenosis | 0-48 hours
  Carotid artery stenosis measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei Wu, MD, Principal Investigator — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided